CLINICAL TRIAL: NCT04157790
Title: Efficacy of the CARE Rule Associated With the HEART Score in Patients With Emergency Chest Pain
Acronym: eCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 49RC19_0071
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-07

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral (No Intervention): Suggested to follow European Society of Cardiology guidelines for NSTEMI
- CARE score (Active Comparator): calculation of the CARE score and prescription for troponins assays or not according to the result (score > 1: troponins assays ; score < 2: no troponins assays)
  Interventions: Other: CARE score

INTERVENTIONS:
Other: CARE score — CARE score calculation
  Arms: CARE score

SUMMARY:
Acute coronary syndrome (ACS) is a major public health problem and its diagnosis remains a challenge for the emergency physician. The European Society of Cardiology recommends a troponin dosage and renew it if necessary during any suspicion of ACS. However, the criteria leading to initiate a diagnostic procedure during chest pain are imprecise. The fear is, on the one hand, to miss a potentially vital diagnosis and, on the other hand, to expose a large number of patients to unnecessary examinations.

The CARE rule (also known as HEAR score) seems to streamline this first step. It assigns a value of 0 to 2 using 4 items: Characteristic of pain, Age, Risk factors and Electrocardiogram (ECG). The search for an ACS is not justified if the sum of the points is <2 (negative rule) and, inversely, a troponin determination must be carried out if the sum is > 1 (positive rule).

The aim of the study is to demonstrate the safety and interest of the CARE rule associated with the HEART score to streamline ACS's diagnostic approach to thoracic pain in emergencies departments.

DETAILED DESCRIPTION:
Data collected in this study are not anticipated to be published in a data repository. However, data will be shared per requested need to researchers, upon presentation of a structured protocol, when approved by the competent ethic committee and approved by the steering committee.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an Emergency Department participating in the study
* Non-traumatic chest pain
* Age greater than or equal to 18 years
* Patient's consent (oral for France, written for Belgium)

Exclusion Criteria:

* 30 days follow-up not possible
* ST-segment Elevation Myocardial Infarction (STEMI) on admittance ECG
* Chest pain formally reported to a diagnosis other than an ACS before inclusion (e.g., pneumothorax, pleurisy, etc.)
* Troponin assay performed prior to inclusion (less than 24 hours old)
* Patient referred by another care structure (excluding primary medicine)
* Patient already included in study still in follow-up period
* Pregnant, breastfeeding or parturient patient,
* Patient deprived of liberty by judicial or administrative decision,
* Patient undergoing psychiatric care under duress,
* Patient subject to a legal protection measure,
* Patient unable to give free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2153 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Rate of major cardiac events | 30 days
  Myocardial infarction, percutaneous or surgical coronary reperfusion, certain or potential cardiac death, or surviving cardiac arrest

SECONDARY OUTCOMES:
Rate of major cardiac events for the intention to treat study population | 30 days
Number of troponin assays in the intention to treat population | 2 days
Time spent in the emergency department in the intention to treat population | 2 days

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU de Liège, Liège
- France (9):
  - CHU Angers, Angers
  - Centre Hospitalier de Cholet, Cholet
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - CH de Saint-Brieuc, Saint-Brieuc
  - CH de Saint-Malo, St-Malo
  - CHU Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Moumneh T, Penaloza A, Charpentier S, Douillet D, Prunier F, Riou J, Roy PM. Efficacy of HEAR and HEART score to rule out major adverse cardiac events in patients presenting to the emergency department with chest pain: study protocol of the eCARE stepped-wedge randomised control trial. BMJ Open. 2022 Dec 6;12(12):e066953. doi: 10.1136/bmjopen-2022-066953. PMID 36600358